CLINICAL TRIAL: NCT02261285
Title: ONO-4538 Multicenter, Open-label, Uncontrolled, Phase I Study in Solid Tumor
Brief Title: ONO-4538 Phase I Study in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-13
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Results first posted 2024-04-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Recurrent Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Increase the dose sequentially.
Oversight: Data Monitoring Committee: No

ARMS (3):
- ONO-4538 1mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 1mg/kg, single dose
  Interventions: Drug: ONO-4538
- ONO-4538 3mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 3mg/kg, single dose
  Interventions: Drug: ONO-4538
- ONO-4538 10mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 10mg/kg, single dose
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538

SUMMARY:
The objective of the study is to investigate the pharmacokinetics of ONO-4538 administered to Korean patients with advanced or recurrent solid tumors who are refractory or intolerant to standard therapy or for whom no appropriate treatment is available.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 years of age
* Histologically or cytologically confirmed solid tumor
* Patients with advanced or recurrent solid tumors who are refractory or intolerant to standard therapy or for whom no appropriate treatment is available
* ECOG Performance Status is 0 to 1

Exclusion Criteria:

* Current or prior severe hypersensitivity to another antibody product
* Multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (5):
- South Korea (5):
  - Seongnam-si Clinical Site 105, Seongnam-si, Gyeonggi-do
  - Seoul Clinical Site 101, Seoul
  - Seoul Clinical Site 102, Seoul
  - Seoul Clinical Site 103, Seoul
  - Seoul Clinical Site 104, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KW, Lee DH, Kang JH, Park JO, Kim SH, Hong YS, Kim ST, Oh DY, Bang YJ. Phase I Pharmacokinetic Study of Nivolumab in Korean Patients with Advanced Solid Tumors. Oncologist. 2018 Feb;23(2):155-e17. doi: 10.1634/theoncologist.2017-0528. Epub 2017 Nov 20. PMID 29158363

RESULTS

PARTICIPANT FLOW:
Groups:
- ONO-4538 1 mg/kg: Subjects with advanced or recurrent solid tumors, received single dose of Nivolumab (ONO-4538) at a dose of 1 mg/kg as an intravenous infusion over approximately 60 minutes.
- ONO-4538 3 mg/kg: Subjects with advanced or recurrent solid tumors, received single dose of Nivolumab (ONO-4538) at a dose of 3 mg/kg as an intravenous infusion over approximately 60 minutes.
- ONO-4538 10 mg/kg: Subjects with advanced or recurrent solid tumors, received single dose of Nivolumab (ONO-4538) at a dose of 10 mg/kg as an intravenous infusion over approximately 60 minutes.
Period: Overall Study
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Started | 6 | 6 | 6
Completed | 6 | 6 | 5
Not Completed | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ONO-4538 1 mg/kg; ONO-4538 3 mg/kg; ONO-4538 10 mg/kg: Refer to "Participant Flow ".
- Total: Total of all reporting groups
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Median (Full Range); unit: years] | 44.5 [36 to 74] | 63.0 [49 to 70] | 52.5 [27 to 84] | 56.0 [27 to 84]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 4 | 3 | 4 | 11
  >=65-<75 years | 2 | 3 | 1 | 6
  >=75 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 4 | 10
  Male | 1 | 5 | 2 | 8
Region of Enrollment [Number; unit: participants]
  South Korea | 6 | 6 | 6 | 18
Height [Median (Full Range); unit: Centimeter] | 156.60 [150.0 to 172.1] | 161.90 [151.0 to 173.0] | 161.35 [157.5 to 174.0] | 160.85 [150.0 to 174.0]
Weight [Median (Full Range); unit: Kilogram] | 56.75 [48.2 to 78.5] | 63.40 [47.0 to 75.0] | 57.50 [49.8 to 68.2] | 59.25 [47.0 to 78.5]
BMI [Median (Full Range); unit: Kilogram per square meter] | 22.62 [19.9 to 28.0] | 23.26 [18.9 to 32.9] | 21.55 [19.3 to 25.8] | 22.57 [18.9 to 32.9]
Performance status (Eastern Cooperative Oncology Group) [Count of Participants; unit: Participants] — PS 0 means "fully active, able to carry on all pre-disease performance without restriction" whereas PS 1 means "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work". Please use the Measure Description to specify how participants were "staged" or "graded" clinically (e.g., briefly describe the criteria for the Rows or Categories) and specify which "stages" or "grades" were considered better or worse outcomes.
  Participants
    PS 0 | 4 | 1 | 3 | 8
    PS 1 | 2 | 5 | 3 | 10
Type of primary cancer [Count of Participants; unit: Participants]
  Lung cancer | 0 | 1 | 3 | 4
  Melanoma | 3 | 0 | 0 | 3
  Salivary gland cancer | 1 | 1 | 0 | 2
  Rectal cancer | 0 | 2 | 0 | 2
  Renal cell carcinoma | 0 | 0 | 1 | 1
  Pancreatic cancer | 0 | 1 | 0 | 1
  Gastric cancer | 1 | 0 | 0 | 1
  Nasal cavity cancer | 0 | 0 | 1 | 1
  Nasopharyngeal carcinoma | 0 | 1 | 0 | 1
  Colon cancer | 0 | 0 | 1 | 1
  Sarcoma | 1 | 0 | 0 | 1
History of surgery [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 3 | 14
  No | 0 | 1 | 3 | 4
History of radiotherapy [Count of Participants; unit: Participants]
  Yes | 4 | 4 | 4 | 12
  No | 2 | 2 | 2 | 6
History of chemotherapy [Count of Participants; unit: Participants]
  None | 1 | 0 | 0 | 1
  1 regimen | 0 | 1 | 1 | 2
  2 regimens | 2 | 1 | 2 | 5
  3 regimens | 1 | 2 | 1 | 4
  4 regimens | 0 | 1 | 2 | 3
  5 regimens | 2 | 0 | 0 | 2
  6 regimens | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: PK Outcome: Cmax of ONO-4538
Description: Cmax was the maximum serum concentration of ONO-4538 after the single administration.
Time Frame: 3 weeks: from the start of administration to the end of treatment phase. Actual blood sampling points are pre-dose, 1hr, 3hr, 9hr, 25hr, 49hr, 73hr, 169hr, 337hr, and 504hr.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
µg/mL | 26.0 (4.29) | 64.3 (22.5) | 242.0 (66.7)

2. Primary Outcome: PK Outcome: Tmax of ONO-4538
Description: Tmax was the time to reach the Cmax.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
hours | 3.02 [1.07 to 9.00] | 3.00 [1.00 to 8.78] | 2.99 [1.00 to 8.62]

3. Primary Outcome: AUC21day
Description: AUC21day was the area under serum concentration-time curve of ONO-4538 from day 0 to day 21 (last measurement).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
µg*h/mL | 5110 (952) | 12200 (2060) | 38700 (14200)

4. Primary Outcome: AUCinf
Description: AUCinf was the area under serum concentration-time curve of ONO-4538 extrapolated to infinity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
µg*h/mL | 9180 (3140) | 22800 (10000) | 68100 (34700)

5. Primary Outcome: T1/2
Description: T1/2 was the elimination half-life of serum concentration of ONO-4538.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
days | 18.3 (6.97) | 19.1 (10.0) | 15.0 (7.86)

6. Secondary Outcome: Safety Outcome: The Number of Subjects With Overall Adverse Events
Description: Adverse Events (AEs) were analyzed based on treatment emergent AEs (TEAEs), defined as any event not present prior to initiation of investigational product that first appeared following exposure to investigational product or any event already present that worsened relative to the pre-treatment state following exposure to investigational product.
Time Frame: 3 weeks: from the start of administration to the end of treatment phase.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants | 5 | 4 | 5

7. Secondary Outcome: Safety Outcome: The Number of Deaths
Description: Number of subjects with TEAEs leading to death.
Time Frame: 3 weeks: from the start of administration to the end of treatment phase.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 weeks: from the start of administration to the end of treatment phase.
Description: Adverse Events (AEs) were analyzed based on treatment emergent AEs (TEAEs), defined as any event not present prior to initiation of investigational product that first appeared following exposure to investigational product or any event already present that worsened relative to the pre-treatment state following the exposure to investigational product. All-Cause Mortality was defined as incidence of subjects who have died during study period.
Arm/Group | ONO-4538 1 mg/kg | ONO-4538 3 mg/kg | ONO-4538 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 1 mg/kg (N=6) | ONO-4538 3 mg/kg (N=6) | ONO-4538 10 mg/kg (N=6)
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 1 mg/kg (N=6) | ONO-4538 3 mg/kg (N=6) | ONO-4538 10 mg/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this tiral prior to submission for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02261285/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02261285/SAP_001.pdf